CLINICAL TRIAL: NCT05084014
Title: EFFECTS OF DEEP STRIPPING VERSUS KNEADING ON PAIN, RANGE OF MOTION AND FUNCTIONAL ACTIVITY AMONG INDIVIDUALS WITH KNEE OSTEOARTHRITIS: A RANDOMIZED CONTROLLED TRIAL
Brief Title: EFFECTS OF DEEP STRIPPING VERSUS KNEADING ON PAIN, RANGE OF MOTION AND FUNCTIONAL ACTIVITY AMONG INDIVIDUALS WITH KNEE OSTEOARTHRITIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/819-I/2021
Record Dates: First submitted 2021-10-03; First posted 2021-10-19 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2024-10

CONDITIONS: Knee Osteoarthritis
Keywords: Non-inflammatory disease; Degenerative joint disease; Osteoarthritis; knee joint; soft tissue mobilization; deep longitudinal stripping; kneading
MeSH Terms: conditions — Osteoarthritis, Knee; Joint Diseases; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: In this study there are two groups, one receiving deep longitudinal stripping technique with conventional physical therapy and the second group receiving kneading technique with conventional physical therapy
Who Masked: Outcomes Assessor
Masking Description: In this study, the outcome assessor will be blinded. He will just take the data regarding pain, functional mobility and measure the range of motion of the knee joint at the baseline, mid of the treatment and at the end of the treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep Stripping (Experimental): This group will receive deep stripping technique with conventional physical therapy.
  Interventions: Other: Deep Stripping
- Kneading (Experimental): This group will receive deep kneading with conventional physical therapy.
  Interventions: Other: Kneading

INTERVENTIONS:
Other: Deep Stripping — The deep longitudinal stripping can be applied on adhesions and knots in muscles. The lengthening stokes are parallel to muscle fiber and applied in an oblique direction with the help of the thumbs of hands/ elbow/ knuckles
  Arms: Deep Stripping
Other: Kneading — kneading lifts the muscle in circular movements with the help of the hands. It lifted, rolled, and squeezed muscle
  Arms: Kneading

SUMMARY:
This is a randomized controlled trial, 44 participants selected based on inclusion criteria from physical therapy department of Surriya Azeem Surgical Hospital, Pattoki. Participants randomly recruited into two groups, 22 in deep stripping group receiving deep stripping with conventional physical therapy and 22 in kneading group receiving kneading with conventional physical therapy. Pain, range of motion and functional mobility are the primary outcomes measured by numeric pain rating scale, universal goniometer and lower extremity functional scale. Data collected at the baseline, at the 6th session, and the 12th session.

DETAILED DESCRIPTION:
In this randomized controlled trial, 44 individuals with knee osteoarthritis (II-III grade of Kellgren-Lawrence scale) pre-diagnosed by an orthopedic, were assessed for eligibility from the physical therapy department of Surriya Azeem Surgical Hospital, Pattoki. Participants with any other musculoskeletal disorder, cognitive problem and receiving any treatment within the past three months were excluded from the study. The participants were randomly recruited into two groups with 22 participants in each group. Group A received deep stripping along with conventional physiotherapy and group B received kneading along with conventional physiotherapy. Both the deep stripping and kneading technique applied on the quadriceps muscle group, hamstring muscle group and around the knee joint. Data collected by a blinded assessor at the baseline, at the 6th session, and the 12th session.

Outcome measures were pain (measured by Numeric Pain Rating Scale), range of motion (measured by Universal Goniometer), and functional mobility (assessed by Lower Extremity Functional Scale). After collecting the data, normality of the data will be entered and analyzed in Statistical Package for the Social Sciences and than the statistical test will be applied to compare the within group analysis and between group analysis.

ELIGIBILITY:
Inclusion Criteria:

* Chronic osteoarthritis (more than 3 months) with pain in one knee joint (unilateral)
* A prior medical diagnosis having radiographic evidence of grade 2 and 3 of Kellgren and Lawrence criteria for knee osteoarthritis by an orthopedic.
* Pain intensity level more than 3 points of the numeric pain rating scale.

Exclusion Criteria:

* Any acute inflammation, contracture, or surgery affecting the knee joint.
* Any cognitive problem.
* Participants taking non-steroid anti-inflammatory drugs, intra-articular injection, or physical therapy within the last three months for the knee joint.
* Participants having a lumbar spine and/or any other lower limb impairment and/or surgery affecting knee joint.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-02-11 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Change from the baseline in Numeric pain rating scale at 2nd and 4th week | Baseline, 2nd week, 4th week
  It is the simplest and most commonly used numeric scale in which the individual rates the pain from 0 (no pain) to 10 (worst pain) 0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7-10 = severe pain
Change from baseline in Universal Goniometer at 2nd and 4th week | Baseline, 2nd week, 4th week
  the range of motion (flexion and extension) measured by using Universal Goniometer. For the range of motion, Universal Goniometer was used. It is an instrument made up of plastic material; it has a moveable arm, stationary arm and a fulcrum. The range of motion of the knee joint in extension and flexion was measured. The normal knee flexion range is 0⁰-130⁰ and the extension range is 130⁰-0⁰.
Change from baseline in Lower Extremity Functional Scale at 2nd and 4th week | Baseline, 2nd week, 4th week
  For functional mobility Lower Extremity Functional Scale is used. This questionnaire contains 20 questions about the ability of a person to carry out his/her daily routine tasks. Every question has 5 options 0 = Extreme difficulty or unable to perform an activity
  1. = Quite a bit of difficulty
  2. = Moderate difficulty
  3. = a little bit of difficulty
  4. = no difficulty. The participant's score was interpreted at the end by adding all the scores of 20 questions, categorizing them into very high function, moderate function, mild function and very low function

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Javed, MSPT-MSK, Principal Investigator — University of Lahore
Locations (1):
- M.Mubeen Javed, Pattoki, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- [Background] Peters AE, Akhtar R, Comerford EJ, Bates KT. The effect of ageing and osteoarthritis on the mechanical properties of cartilage and bone in the human knee joint. Sci Rep. 2018 Apr 12;8(1):5931. doi: 10.1038/s41598-018-24258-6. PMID 29651151
- [Background] Ilas DC, Churchman SM, McGonagle D, Jones E. Targeting subchondral bone mesenchymal stem cell activities for intrinsic joint repair in osteoarthritis. Future Sci OA. 2017 Sep 6;3(4):FSO228. doi: 10.4155/fsoa-2017-0055. eCollection 2017 Nov. PMID 29134116
- [Background] Karaborklu Argut S, Celik D, Kilicoglu OI. The Combination of Exercise and Manual Therapy Versus Exercise Alone in Total Knee Arthroplasty Rehabilitation: A Randomized Controlled Clinical Trial. PM R. 2021 Oct;13(10):1069-1078. doi: 10.1002/pmrj.12542. Epub 2021 Feb 3. PMID 33352007
- [Background] Ferreira RM, Torres RT, Duarte JA, Goncalves RS. Non-Pharmacological and Non-Surgical Interventions for Knee Osteoarthritis: A Systematic Review and Meta-Analysis. Acta Reumatol Port. 2019 Jul 29;44(3):173-217. PMID 31356585
- [Background] Perlman A, Fogerite SG, Glass O, Bechard E, Ali A, Njike VY, Pieper C, Dmitrieva NO, Luciano A, Rosenberger L, Keever T, Milak C, Finkelstein EA, Mahon G, Campanile G, Cotter A, Katz DL. Efficacy and Safety of Massage for Osteoarthritis of the Knee: a Randomized Clinical Trial. J Gen Intern Med. 2019 Mar;34(3):379-386. doi: 10.1007/s11606-018-4763-5. Epub 2018 Dec 12. PMID 30543021